CLINICAL TRIAL: NCT03043781
Title: The Programmed Intermittent Epidural Bolus Adrenaline Study
Acronym: PIEBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Vegard Dahl, Principal investigator, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-004397-14
Record Dates: First submitted 2017-01-31; First posted 2017-02-06 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermittent epidural bolus (IEB) (Experimental): Bolus of 5 ml every hour + patient controlled extra boluses of 5 ml, maximum 3 / hour. Medicine solution is bupivacaine 1 mg/ml, fentanyl 2 mcg/ml, adrenaline 2 mcg/ml.
  Interventions: Other: Intermittent epidural bolus
- Continuous epidural infusion (CEI) (Active Comparator): Continuous epidural infusion of 5 ml / hour + patient controlled extra boluses of 5 ml, maximum 3 / hour. Medicine solution is bupivacaine 1 mg/ml, fentanyl 2 mcg/ml, adrenaline 2 mcg/ml.
  Interventions: Other: Continuous epidural infusion

INTERVENTIONS:
Other: Continuous epidural infusion — Continuous infusion, 5 ml/h
  Arms: Continuous epidural infusion (CEI)
Other: Intermittent epidural bolus — Intermittent bolus 5 ml every hour
  Arms: Intermittent epidural bolus (IEB)

SUMMARY:
This study evaluates the use of intermittent epidural boluses compared to continuous infusion in maintaining epidural pain relief in labor.

The medicine solution used contains, in addition to bupivacain and fentanyl, adrenalin in both groups.

DETAILED DESCRIPTION:
Labor is often painful for the woman going through it, and thus many women choose to have pain relief by an epidural catheter.

This is done by placing a thin plastic catheter in the epidural space in the lower back of the patient, and injecting a medicine solution usually consisting of local anesthesia and opioids.

To ensure an effective pain relief through the labor process, additional medicine solution is injected through the catheter. Traditionally, this is done by a continuous infusion, often with the addition of patient controlled boluses.

In this study the investigators investigate if maintaining the pain relief through programmed hourly intermittent boluses is more effective than continuous infusion. This is done in other studies with promising results, but the difference in this study is the addition of adrenaline to the medicine solution in order to make it more effective.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in labor requesting epidural analgesia
* ASA group 1 and 2
* 0 or 1 previous births
* Must be at least 18 years of age.
* Singleton pregnancy
* Active labor
* Signed informed consent and expected cooperation of the patient

Exclusion Criteria:

* Poor communication skills in norwegian or english
* Adverse reactions to local anesthetics or synthetic opioids
* Body height below 150 cm
* Gestational age below 37 weeks, 0 days
* Any contraindication to epidural catheter placement (e.g. patients with coagulopathy, infection in area etc)
* Pre-eclampsia
* Sound reason by the investigator to suspect patient non-compliance (e.g. with use of PCEA)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Cumulative drug consumption, time adjusted | One assessment, within 24 hours of end of treatment
  Cumulative drug consumption is assessed at the end of treatment (at birth). The total dose is adjusted for differences in treatment time and other possible factors of influence (BMI, parity, age, gestational age etc.)

SECONDARY OUTCOMES:
Maternal satisfaction with treatment | One assessment, within 24 hours of end of treatment
  Overall satisfaction with treatment will be assessed the day after end of treatment on a 0-10 scale.
Mode of delivery | One assessment, within 24 hours of end of treatment
  Mode of delivery will be assessed and categorized as vaginal,instrumentally assisted or cesarean delivery.
Motor block | One assessment at one hour after treatment initiation and one at 10 cm cervical dilatation.
  Extent of lower extremity motor block will be assessed using a modified Bromage score
Anesthesiologic intervention | During treatment (0-24 hours)
  The need for additional anesthesiologic intervention, including time to this intervention from start of treatment.
Incidence of expected adverse events | Adverse events during treatment (0-24 hours) and final assessment within 24 hours of end of treatment
  Expected adverse events include hypotension (systolic blood pressure < 90 mmHg and/or use of vasopressors), nausea (mild/moderate/severe) and pruritus (mild/moderate/severe).
Pain rating | During treatment (0-24 hours)
  Pain rating will be assessed using a numeric rating scale (NRS, 0-10; 0= no pain, 10=worst imaginable pain) before treatment start, at every hour for the first 8 hours of treatment and every other hour thereafter. Worst pain at delivery will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Dahl, MD, Dr. Med., Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus UH, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data.

REFERENCES:
- [Background] George RB, Allen TK, Habib AS. Intermittent epidural bolus compared with continuous epidural infusions for labor analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jan;116(1):133-44. doi: 10.1213/ANE.0b013e3182713b26. Epub 2012 Dec 7. PMID 23223119